CLINICAL TRIAL: NCT05763212
Title: Effects Of Reverse Walking With And Without Whole Body Vibration On Postural Balance And Quality Of Life In Children With Cerebral Palsy
Brief Title: Reverse Walking With And Without Whole Body Vibration in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0739
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Cerebral Palsy
Keywords: postural balance
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reverse Walking+Baseline treatment (Active Comparator): Conventional treatment was given then received Reverse Walking Training which was provided for 7 min per set, with approximately 3 min of inter-set rest, for a total training duration of 60 min/day, 3 days/week for 3 successive months .
  Interventions: Other: Reverse Walking+Baseline treatment
- Whole Body Vibration + Reverse Walking+Baseline treatment (Experimental): Conventional Physical Therapy Treatment was given as a baseline treatment which includes Stretching, Range of motion exercises, and Strengthening exercises) performed for 10 min.
  Reverse Walking Training which was provided for 7 min per set, with approximately 3 min of inter-set rest, for a total training duration of 30 min/day, 3 days/week for 3 successive months After that Group received Whole Body Vibration including three vibration sessions per week for three months. The participants have to carry out each set of vibration for 2 min in the first month, and then it was increased to 3 min in the second and 5 min in the third month. The rest period between each set was 1 min in the first month, then it became half a minute in the second and third month. Total training duration is 30 min/day, 3 days/week for 3 successive months.
  Interventions: Other: Whole Body Vibration + Reverse Walking+Baseline treatment

INTERVENTIONS:
Other: Reverse Walking+Baseline treatment — Reverse Walking+Baseline treatment
  Arms: Reverse Walking+Baseline treatment
Other: Whole Body Vibration + Reverse Walking+Baseline treatment — Whole Body Vibration + Reverse Walking+Baseline treatment
  Arms: Whole Body Vibration + Reverse Walking+Baseline treatment

SUMMARY:
To determine the effects of reverse walking with and without Whole-body vibration on postural balance in children with cerebral palsy.

DETAILED DESCRIPTION:
Current study concluded that reverse walking with and without whole body vibration were effective in improving postural balance, reach and quality of life in cerebral palsy children. However (whole body vibration+ reverse walking) provides more clinical benefits than reverse walking alone in improving postural balance, side reach and quality of life. Whereas both techniques were equally effective in improving forward reach in cerebral palsy children.

ELIGIBILITY:
Inclusion Criteria:

Aged 6-12 years

* Confirm diagnosis of Cerebral Palsy
* GMFCS level I & II
* Both genders (28)

Exclusion Criteria:

* o Visual impairment

  * Patients who can't follow command
  * Hearing impairment
  * Malignancy
  * Infection (such as Osteomyelitis)
  * Inflammatory arthritis
  * Lower extremity bones fracture
  * Cardiovascular disease
  * Traumatic cases

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale; | 12th week
  The pediatric balance scale is the modified version of the berg balance scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points
Pediatric Reach Test (PRT) / Functional Reach Test (FRT) | 12th week
  The Pediatric Reach Test (PRT) is a modified form of the Functional Reach Test (FRT). The PRT measures side reaching as well as forward reaching in both sitting and standing positions.

SECONDARY OUTCOMES:
CP QOL-Child | 12th week
  The CP QOL-Child was designed to assess the quality of life of children aged 4-12 years. There are two versions, including a primary caregiver/parent report for children aged 4 to 12 years; and a self-report for children aged 9 to 12 years(10).
  GMFCS level I & II GMFCS Level I

CONTACTS AND LOCATIONS:
Overall Officials: fareeha kausar, pp-Dpt, Principal Investigator — Riphah international university pakistan
Locations (1):
- Hussain memorial hospital lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No